CLINICAL TRIAL: NCT05067777
Title: Massage for Prostate Cancer-Related Fatigue (mPROSTATE)
Acronym: mPROSTATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCI144295; NCI-2021-09613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI144295 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH); R21CA263453 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-10-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Massage

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Swedish Massage Therapy (SMT) (Experimental): Patients receive SMT over 45 minutes once weekly for 6 weeks.
  Interventions: Procedure: Swedish Massage Therapy (SMT)
- Light Touch (LT) (Sham Comparator): Patients receive LT over 45 minutes once weekly for 6 weeks.
  Interventions: Procedure: Light Touch (LT) Control
- Waitlist Control (WLC) (Active Comparator): Patients will sit and relax for 45 minutes before completing study assessments at weeks 3 and 6.
  Interventions: Other: Waitlist Control (WLC)

INTERVENTIONS:
Procedure: Swedish Massage Therapy (SMT) — The therapist uses non-aromatic cream to facilitate making long strokes over the body. Swedish massage is done with the subject covered by a sheet, a technique called "draping." One part of the body is uncovered, massaged, and then re-draped before moving to another part. The primary techniques used in the research protocol therapy are effleurage, petrissage, kneading, tapotement and thumb friction. These techniques are performed in a very precise, carefully elaborated manner. The session starts with the subject fully draped in a prone position on the massage table and after approximately 22 minutes the subject is instructed to turn to the supine position. Finally, the therapist moves to the head area of the subject, begins working on the shoulders, neck and head using effleurage and thumb friction, and concludes by using light tapotement on the head. The total time for the entire massage is 45 minutes.
  Other Names: Massage; massage therapy
  Arms: Swedish Massage Therapy (SMT)
Procedure: Light Touch (LT) Control — The protocol entails the same duration and sequence of procedures as the massage protocol, except that the therapist employs only light-touch hand placement on the subject's body. This condition isolates the effect of the mechanical intervention of SMT.
  Arms: Light Touch (LT)
Other: Waitlist Control (WLC) — Subjects randomized to WLC will sit and relax for 45 minutes.
  Other Names: Sham Intervention
  Arms: Waitlist Control (WLC)

SUMMARY:
This phase II trial investigates the effect of massage in decreasing prostate cancer-related fatigue. Massage therapy has well known health benefits. This trial aims to find out if massage and touch therapies reduce fatigue due to cancer, and to learn if these therapies are better than traditional medicine or psychology for cancer related fatigue.

DETAILED DESCRIPTION:
With over 15.5 million cancer survivors today in the United States, increased attention is being given to quality of life (QOL) after cancer treatment. Cancer-related fatigue (CRF), "a persistent, subjective sense of physical, emotional, and/or cognitive exhaustion related to cancer or its treatment that is not proportional to recent activity" (National Comprehensive Cancer Network, accessed Oct2020), is the most common and one of the most devastating symptoms among patients with cancer. CRF occurs across the spectrum of cancer types and treatments and has a negative impact on all areas of function, including mood, physical function, work performance, social interaction, family care, cognitive performance, schoolwork, and community activities. CRF can persist for months or years after cancer therapy is completed. CRF has been designated a high-priority research area by the National Cancer Institute (NCI) and is 1 of the 5 highest-priority research areas designated by the NCI Clinical Oncology Research.

This study is a phase II, 3-arm, randomized comparison of single-blinded once-weekly Swedish Massage Therapy (SMT) vs. Light Touch (LT) Control vs. unblinded waitlist control (WLC) for 6 weeks. We chose once-a-week sessions for 6 weeks to match the length of our completed National Center for Complementary and Integrative Health (NCCIH) trial of SMT vs. LT for breast cancer survivors with CRF.

Subjects who complete SMT or LT will be interviewed in person, by telemedicine, or by telephone at 6 and 12 weeks after the last study visit in order to evaluate the sustained effects of SMT and LT. We hypothesize that SMT will have a clinically meaningful benefit in improving fatigue, mood, and quality of life (QOL) in Prostate Cancer (PCa) patients, and that this will correlate with favorable changes in physiological parameters that may underlie CRF. Demographic, medical, clinical, and biological characteristics will be compared between groups of subjects randomized to SMT, LT, or WLC. Any treatment group differences in PCa grade and time since completion of radiation therapy, or baseline Brief Fatigue Inventory (BFI) fatigue score, may affect treatment-related change in fatigue or biological measures related to inflammation, or the post-treatment duration of benefit. While groups are expected to be similar on these characteristics, any variable with a p ≤ 0.10 difference between groups will be considered as a candidate covariate or stratification variable for statistical tests of the study hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged >= 45 years old
* Histologically confirmed diagnosis of prostate cancer
* Subjects must have completed radiation therapy >= 2 months, prior to registration
* Subjects who have a score > 25 on the Brief Fatigue Inventory (BFI) at screening
* Subjects who are fluent in speaking and reading English
* Based on International Classification of Diseases (ICD)-10 proposed criteria, the patient must have a diagnosis of CRF with evidence from the history, physical exam, and laboratory findings that the fatigue is a consequence of cancer or cancer therapy and not primarily a consequence of any of the following:

  * Comorbid psychiatric disorders
  * Anemia (hemoglobin less than 10 g/dl)
  * Hypothyroidism (thyroid stimulating hormone (TSH) greater than 4.6 micro-international units (uIU)/mL)
  * Uncontrolled pain
  * Any medical or psychiatric condition or medication felt to be clinically contributing to fatigue based on the investigator's history, physical examination, and assessment. These medical circumstances may include:

    * The use of medications such as opioids, sedating anti-histamines, or neuroleptics;
    * Medical problems associated with fatigue: chronic obstructive pulmonary disease, congestive heart failure, renal disease, hepatic dysfunction, uncontrolled autoimmune disease, neurological disorders such as multiple sclerosis or Parkinson's disease, and sleep apnea
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Inability to lay prone comfortably for 25 minutes and inability to lay supine comfortably for 25 minutes, given the nature of the massage intervention
* Body-mass index less than 18.5 (kg/m^2)
* Current use of any medications or therapies listed as prohibited in Section 6.6.1.
* Treatment with corticosteroids or other immunosuppressants =< 6 months prior to registration, , unless the medication is necessary to support patient wellbeing and unlikely to negatively impact study aims, per PI judgement..
* Subjects who cannot comply with the protocol for any reason
* Regular use of anti-inflammatory drugs including non-steroidal anti-inflammatory drugs and natural products thought to have anti-inflammatory properties, unless the medication is necessary to support patient wellbeing and unlikely to negatively impact study aims, per PI judgement.
* Change in prescribed dose of medications for anxiety or depression =< 4 weeks prior to registration.
* Change in fluoxetine dose within =< 8 weeks prior to registration
* Subjects meeting criteria for a current substance use diagnosis or current diagnoses of schizophrenia, depression, generalized anxiety disorder, bipolar disorder, dementia, delirium, or obsessive compulsive disorder (OCD)
* Subjects who are actively suicidal or homicidal
* Other conditions or behaviors that, in the opinion of the treating investigator, may negatively impact study participation, including the following:

  * Illicit drug use
  * Shift work
  * Current dieting
  * Excessive regular use of alcohol (more than two 5-ounce glasses of wine or equivalents/day)
  * Any instance of binge drinking (more than 7 drinks in a 24-hour period) =< 6 months prior to registration
* Current and/or past use of massage for the treatment of fatigue.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol, or complete the study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Change in cancer-related fatigue | up to 6 weeks from the initiation of study intervention
  Multidimensional Fatigue Inventory (MFI)-20 is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Participants rate each item on a 5-point Likert scale from 1 "yes, that is true" to 5 "no, that is not true".
  This outcome measure will report 5 subscales (General Fatigue, Physical Fatigue, Reduced Activity, Reduced Motivation, Mental Fatigue) and the Total Raw Score. All scores range from 1-5, with higher scores indicating more fatigue and lower scores indicating less fatigue.

SECONDARY OUTCOMES:
Change in plasma concentrations of pre-inflammatory cytokine IL-1beta | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine IL-1beta from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in IL-1beta and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine IL-1Ra | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine IL-1Ra from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine IL-1Ra and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine IL-6 | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine IL-6 from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine IL-6 and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine sIL-6R | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine sIL-6R from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine sIL-6R and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine TNF-α | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine TNF-α from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine TNF-α and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine sTNFR2 | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine sTNFR2 from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine sTNFR2 and MFI scores.
Change in plasma concentrations of pre-inflammatory cytokine IFN-γ | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of pre-inflammatory cytokine IFN-γ from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in cytokine IFN-γ and MFI scores.
Change in plasma concentrations of High-Sensitivity C-Reactive Protein (hsCRP) | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of hsCRP from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in hsCRP and MFI scores.
Change in plasma concentrations of anti-inflammatory cytokine IL-10 | up to 6 weeks from the initiation of study intervention
  To evaluate whether the hypothesized decrease in cancer-related fatigue with SMT is associated with modulation of specific immune system factors underlying chronic inflammation.
  This outcome measure will report the mean change in plasma concentrations of anti-inflammatory cytokine IL-10 from baseline to 6 weeks after initiation of the study intervention.
  Further statistical analysis will assess the association between the change in anti-inflammatory cytokine IL-10 and MFI scores.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Rapaport, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Curt GA, Breitbart W, Cella D, Groopman JE, Horning SJ, Itri LM, Johnson DH, Miaskowski C, Scherr SL, Portenoy RK, Vogelzang NJ. Impact of cancer-related fatigue on the lives of patients: new findings from the Fatigue Coalition. Oncologist. 2000;5(5):353-60. doi: 10.1634/theoncologist.5-5-353. PMID 11040270
- [Background] Hofman M, Ryan JL, Figueroa-Moseley CD, Jean-Pierre P, Morrow GR. Cancer-related fatigue: the scale of the problem. Oncologist. 2007;12 Suppl 1:4-10. doi: 10.1634/theoncologist.12-S1-4. PMID 17573451
- [Background] Lawrence DP, Kupelnick B, Miller K, Devine D, Lau J. Evidence report on the occurrence, assessment, and treatment of fatigue in cancer patients. J Natl Cancer Inst Monogr. 2004;(32):40-50. doi: 10.1093/jncimonographs/lgh027. PMID 15263040
- [Background] Mehnert A, Hartung TJ, Friedrich M, Vehling S, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Weis J, Koch U, Faller H. One in two cancer patients is significantly distressed: Prevalence and indicators of distress. Psychooncology. 2018 Jan;27(1):75-82. doi: 10.1002/pon.4464. Epub 2017 Jun 16. PMID 28568377
- [Background] Ma Y, He B, Jiang M, Yang Y, Wang C, Huang C, Han L. Prevalence and risk factors of cancer-related fatigue: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Nov;111:103707. doi: 10.1016/j.ijnurstu.2020.103707. Epub 2020 Jul 11. PMID 32920423
- [Background] National Coalition for Cancer Survivorship. Cancer survivorship survey: findings from an online survey of adult cancer patients. https://www.canceradvocacy.org/wpcontent/uploads/2019/09/NCCS-Survivorship-Survey-Final-Report.pdf. , 2019
- [Background] Nail LM. My get up and go got up and went: fatigue in people with cancer. J Natl Cancer Inst Monogr. 2004;(32):72-5. doi: 10.1093/jncimonographs/lgh021. PMID 15263043
- [Background] Berger AM, Kuhn BR, Farr LA, Von Essen SG, Chamberlain J, Lynch JC, Agrawal S. One-year outcomes of a behavioral therapy intervention trial on sleep quality and cancer-related fatigue. J Clin Oncol. 2009 Dec 10;27(35):6033-40. doi: 10.1200/JCO.2008.20.8306. Epub 2009 Nov 2. PMID 19884558
- [Background] Bower JE. Prevalence and causes of fatigue after cancer treatment: the next generation of research. J Clin Oncol. 2005 Nov 20;23(33):8280-2. doi: 10.1200/JCO.2005.08.008. Epub 2005 Oct 11. No abstract available. PMID 16219929
- [Background] Berger AM, Mooney K, Alvarez-Perez A, Breitbart WS, Carpenter KM, Cella D, Cleeland C, Dotan E, Eisenberger MA, Escalante CP, Jacobsen PB, Jankowski C, LeBlanc T, Ligibel JA, Loggers ET, Mandrell B, Murphy BA, Palesh O, Pirl WF, Plaxe SC, Riba MB, Rugo HS, Salvador C, Wagner LI, Wagner-Johnston ND, Zachariah FJ, Bergman MA, Smith C; National comprehensive cancer network. Cancer-Related Fatigue, Version 2.2015. J Natl Compr Canc Netw. 2015 Aug;13(8):1012-39. doi: 10.6004/jnccn.2015.0122. PMID 26285247
- [Background] Boelhouwer IG, Vermeer W, van Vuuren T. The associations between late effects of cancer treatment, work ability and job resources: a systematic review. Int Arch Occup Environ Health. 2021 Feb;94(2):147-189. doi: 10.1007/s00420-020-01567-w. Epub 2020 Sep 15. PMID 32929528
- [Background] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Background] Curran SL, Beacham AO, Andrykowski MA. Ecological momentary assessment of fatigue following breast cancer treatment. J Behav Med. 2004 Oct;27(5):425-44. doi: 10.1023/b:jobm.0000047608.03692.0c. PMID 15675633
- [Background] Committee N-SMQoLS: Strategic Priorities. https://www.cancer.gov/aboutnci/organization/ccct/steering-committees/2015-sxqolsc-strategicpriorities Accessed 10-2020., 2015
- [Background] Ebede CC, Jang Y, Escalante CP. Cancer-Related Fatigue in Cancer Survivorship. Med Clin North Am. 2017 Nov;101(6):1085-1097. doi: 10.1016/j.mcna.2017.06.007. Epub 2017 Aug 25. PMID 28992856
- [Background] Thong MSY, van Noorden CJF, Steindorf K, Arndt V. Cancer-Related Fatigue: Causes and Current Treatment Options. Curr Treat Options Oncol. 2020 Feb 5;21(2):17. doi: 10.1007/s11864-020-0707-5. PMID 32025928
- [Background] Alexander S, Minton O, Andrews P, Stone P. A comparison of the characteristics of disease-free breast cancer survivors with or without cancer-related fatigue syndrome. Eur J Cancer. 2009 Feb;45(3):384-92. doi: 10.1016/j.ejca.2008.09.010. Epub 2008 Oct 30. PMID 18977131
- [Background] Barsevick A, Frost M, Zwinderman A, Hall P, Halyard M; GENEQOL Consortium. I'm so tired: biological and genetic mechanisms of cancer-related fatigue. Qual Life Res. 2010 Dec;19(10):1419-27. doi: 10.1007/s11136-010-9757-7. Epub 2010 Oct 16. PMID 20953908
- [Background] Ryan JL, Carroll JK, Ryan EP, Mustian KM, Fiscella K, Morrow GR. Mechanisms of cancer-related fatigue. Oncologist. 2007;12 Suppl 1:22-34. doi: 10.1634/theoncologist.12-S1-22. PMID 17573453
- [Background] Morrow GR, Andrews PL, Hickok JT, Roscoe JA, Matteson S. Fatigue associated with cancer and its treatment. Support Care Cancer. 2002 Jul;10(5):389-98. doi: 10.1007/s005200100293. Epub 2001 Aug 15. PMID 12136222
- [Background] Roscoe JA, Morrow GR, Hickok JT, Bushunow P, Matteson S, Rakita D, Andrews PL. Temporal interrelationships among fatigue, circadian rhythm and depression in breast cancer patients undergoing chemotherapy treatment. Support Care Cancer. 2002 May;10(4):329-36. doi: 10.1007/s00520-001-0317-0. Epub 2001 Nov 28. PMID 12029433
- [Background] MacHale SM, Cavanagh JT, Bennie J, Carroll S, Goodwin GM, Lawrie SM. Diurnal variation of adrenocortical activity in chronic fatigue syndrome. Neuropsychobiology. 1998 Nov;38(4):213-7. doi: 10.1159/000026543. PMID 9813459
- [Background] Bower JE, Ganz PA, Dickerson SS, Petersen L, Aziz N, Fahey JL. Diurnal cortisol rhythm and fatigue in breast cancer survivors. Psychoneuroendocrinology. 2005 Jan;30(1):92-100. doi: 10.1016/j.psyneuen.2004.06.003. PMID 15358446
- [Background] Bower JE, Ganz PA, Aziz N. Altered cortisol response to psychologic stress in breast cancer survivors with persistent fatigue. Psychosom Med. 2005 Mar-Apr;67(2):277-80. doi: 10.1097/01.psy.0000155666.55034.c6. PMID 15784794
- [Background] Bower JE, Ganz PA, Aziz N, Fahey JL. Fatigue and proinflammatory cytokine activity in breast cancer survivors. Psychosom Med. 2002 Jul-Aug;64(4):604-11. doi: 10.1097/00006842-200207000-00010. PMID 12140350
- [Background] Schrepf A, Clevenger L, Christensen D, DeGeest K, Bender D, Ahmed A, Goodheart MJ, Dahmoush L, Penedo F, Lucci JA 3rd, Ganjei-Azar P, Mendez L, Markon K, Lubaroff DM, Thaker PH, Slavich GM, Sood AK, Lutgendorf SK. Cortisol and inflammatory processes in ovarian cancer patients following primary treatment: relationships with depression, fatigue, and disability. Brain Behav Immun. 2013 Mar;30 Suppl(0):S126-34. doi: 10.1016/j.bbi.2012.07.022. Epub 2012 Aug 5. PMID 22884960
- [Background] Saligan LN, Kim HS. A systematic review of the association between immunogenomic markers and cancer-related fatigue. Brain Behav Immun. 2012 Aug;26(6):830-48. doi: 10.1016/j.bbi.2012.05.004. Epub 2012 May 14. PMID 22595751
- [Background] Wright F, Hammer M, Paul SM, Aouizerat BE, Kober KM, Conley YP, Cooper BA, Dunn LB, Levine JD, DEramo Melkus G, Miaskowski C. Inflammatory pathway genes associated with inter-individual variability in the trajectories of morning and evening fatigue in patients receiving chemotherapy. Cytokine. 2017 Mar;91:187-210. doi: 10.1016/j.cyto.2016.12.023. Epub 2017 Jan 19. PMID 28110208
- [Background] Reyes-Gibby CC, Wu X, Spitz M, Kurzrock R, Fisch M, Bruera E, Shete S. Molecular epidemiology, cancer-related symptoms, and cytokines pathway. Lancet Oncol. 2008 Aug;9(8):777-85. doi: 10.1016/S1470-2045(08)70197-9. PMID 18672213
- [Background] Santos JC, Pyter LM. Neuroimmunology of Behavioral Comorbidities Associated With Cancer and Cancer Treatments. Front Immunol. 2018 Jun 7;9:1195. doi: 10.3389/fimmu.2018.01195. eCollection 2018. PMID 29930550
- [Background] Haroon E, Miller AH. Inflammation Effects on Brain Glutamate in Depression: Mechanistic Considerations and Treatment Implications. Curr Top Behav Neurosci. 2017;31:173-198. doi: 10.1007/7854_2016_40. PMID 27830574
- [Background] Miller AH, Haroon E, Felger JC. Therapeutic Implications of Brain-Immune Interactions: Treatment in Translation. Neuropsychopharmacology. 2017 Jan;42(1):334-359. doi: 10.1038/npp.2016.167. Epub 2016 Aug 24. PMID 27555382
- [Background] Felger JC, Li Z, Haroon E, Woolwine BJ, Jung MY, Hu X, Miller AH. Inflammation is associated with decreased functional connectivity within corticostriatal reward circuitry in depression. Mol Psychiatry. 2016 Oct;21(10):1358-65. doi: 10.1038/mp.2015.168. Epub 2015 Nov 10. PMID 26552591
- [Background] Goldsmith DR, Haroon E, Woolwine BJ, Jung MY, Wommack EC, Harvey PD, Treadway MT, Felger JC, Miller AH. Inflammatory markers are associated with decreased psychomotor speed in patients with major depressive disorder. Brain Behav Immun. 2016 Aug;56:281-8. doi: 10.1016/j.bbi.2016.03.025. Epub 2016 Apr 1. PMID 27040122
- [Background] Irwin MR, Opp MR. Sleep Health: Reciprocal Regulation of Sleep and Innate Immunity. Neuropsychopharmacology. 2017 Jan;42(1):129-155. doi: 10.1038/npp.2016.148. Epub 2016 Aug 11. PMID 27510422
- [Background] Irwin MR, Olmstead R, Carroll JE. Sleep Disturbance, Sleep Duration, and Inflammation: A Systematic Review and Meta-Analysis of Cohort Studies and Experimental Sleep Deprivation. Biol Psychiatry. 2016 Jul 1;80(1):40-52. doi: 10.1016/j.biopsych.2015.05.014. Epub 2015 Jun 1. PMID 26140821
- [Background] Bower JE, Ganz PA, Irwin MR, Castellon S, Arevalo J, Cole SW. Cytokine genetic variations and fatigue among patients with breast cancer. J Clin Oncol. 2013 May 1;31(13):1656-61. doi: 10.1200/JCO.2012.46.2143. Epub 2013 Mar 25. PMID 23530106
- [Background] Smith AK, Conneely KN, Pace TW, Mister D, Felger JC, Kilaru V, Akel MJ, Vertino PM, Miller AH, Torres MA. Epigenetic changes associated with inflammation in breast cancer patients treated with chemotherapy. Brain Behav Immun. 2014 May;38:227-36. doi: 10.1016/j.bbi.2014.02.010. Epub 2014 Feb 28. PMID 24583204
- [Background] Bower JE, Lamkin DM. Inflammation and cancer-related fatigue: mechanisms, contributing factors, and treatment implications. Brain Behav Immun. 2013 Mar;30 Suppl(0):S48-57. doi: 10.1016/j.bbi.2012.06.011. Epub 2012 Jul 6. PMID 22776268
- [Background] LaVoy EC, Fagundes CP, Dantzer R. Exercise, inflammation, and fatigue in cancer survivors. Exerc Immunol Rev. 2016;22:82-93. PMID 26853557
- [Background] Collado-Hidalgo A, Bower JE, Ganz PA, Cole SW, Irwin MR. Inflammatory biomarkers for persistent fatigue in breast cancer survivors. Clin Cancer Res. 2006 May 1;12(9):2759-66. doi: 10.1158/1078-0432.CCR-05-2398. PMID 16675568
- [Background] Paulsen O, Laird B, Aass N, Lea T, Fayers P, Kaasa S, Klepstad P. The relationship between pro-inflammatory cytokines and pain, appetite and fatigue in patients with advanced cancer. PLoS One. 2017 May 25;12(5):e0177620. doi: 10.1371/journal.pone.0177620. eCollection 2017. PMID 28542626
- [Background] Lacourt TE, Vichaya EG, Escalante C, Manzullo EF, Gunn B, Hess KR, Heijnen CJ, Dantzer R. An effort expenditure perspective on cancer-related fatigue. Psychoneuroendocrinology. 2018 Oct;96:109-117. doi: 10.1016/j.psyneuen.2018.06.009. Epub 2018 Jun 9. PMID 29929087
- [Background] Berger AM, Mitchell SA, Jacobsen PB, Pirl WF. Screening, evaluation, and management of cancer-related fatigue: Ready for implementation to practice? CA Cancer J Clin. 2015 May-Jun;65(3):190-211. doi: 10.3322/caac.21268. Epub 2015 Mar 11. PMID 25760293
- [Background] Bruera E, Yennurajalingam S. Challenge of managing cancer-related fatigue. J Clin Oncol. 2010 Aug 10;28(23):3671-2. doi: 10.1200/JCO.2010.29.8984. Epub 2010 Jul 12. No abstract available. PMID 20625135
- [Background] Pachman DR, Price KA, Carey EC. Nonpharmacologic approach to fatigue in patients with cancer. Cancer J. 2014 Sep-Oct;20(5):313-8. doi: 10.1097/PPO.0000000000000064. PMID 25299140
- [Background] Minton O, Stone P, Richardson A, Sharpe M, Hotopf M. Drug therapy for the management of cancer related fatigue. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD006704. doi: 10.1002/14651858.CD006704.pub2. PMID 18254112
- [Background] Vapiwala N, Mick R, Hampshire MK, Metz JM, DeNittis AS. Patient initiation of complementary and alternative medical therapies (CAM) following cancer diagnosis. Cancer J. 2006 Nov-Dec;12(6):467-74. doi: 10.1097/00130404-200611000-00006. PMID 17207316
- [Background] Calcagni N, Gana K, Quintard B. A systematic review of complementary and alternative medicine in oncology: Psychological and physical effects of manipulative and body-based practices. PLoS One. 2019 Oct 17;14(10):e0223564. doi: 10.1371/journal.pone.0223564. eCollection 2019. PMID 31622362
- [Background] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Background] Scott K, Posmontier B. Exercise Interventions to Reduce Cancer-Related Fatigue and Improve Health-Related Quality of Life in Cancer Patients. Holist Nurs Pract. 2017 Mar/Apr;31(2):66-79. doi: 10.1097/HNP.0000000000000194. PMID 28181972
- [Background] Mustian KM, Cole CL, Lin PJ, Asare M, Fung C, Janelsins MC, Kamen CS, Peppone LJ, Magnuson A. Exercise Recommendations for the Management of Symptoms Clusters Resulting From Cancer and Cancer Treatments. Semin Oncol Nurs. 2016 Nov;32(4):383-393. doi: 10.1016/j.soncn.2016.09.002. Epub 2016 Oct 21. PMID 27776835
- [Background] Puetz TW, Herring MP. Differential effects of exercise on cancer-related fatigue during and following treatment: a meta-analysis. Am J Prev Med. 2012 Aug;43(2):e1-24. doi: 10.1016/j.amepre.2012.04.027. PMID 22813691
- [Background] Hilfiker R, Meichtry A, Eicher M, Nilsson Balfe L, Knols RH, Verra ML, Taeymans J. Exercise and other non-pharmaceutical interventions for cancer-related fatigue in patients during or after cancer treatment: a systematic review incorporating an indirect-comparisons meta-analysis. Br J Sports Med. 2018 May;52(10):651-658. doi: 10.1136/bjsports-2016-096422. Epub 2017 May 13. PMID 28501804
- [Background] Kelley GA, Kelley KS. Exercise and cancer-related fatigue in adults: a systematic review of previous systematic reviews with meta-analyses. BMC Cancer. 2017 Oct 23;17(1):693. doi: 10.1186/s12885-017-3687-5. PMID 29058631
- [Background] Chen YJ, Li XX, Ma HK, Zhang X, Wang BW, Guo TT, Xiao Y, Bing ZT, Ge L, Yang KH, Han XM. Exercise Training for Improving Patient-Reported Outcomes in Patients With Advanced-Stage Cancer: A Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2020 Mar;59(3):734-749.e10. doi: 10.1016/j.jpainsymman.2019.09.010. Epub 2019 Sep 20. PMID 31546002
- [Background] Bower JE, Garet D, Sternlieb B, Ganz PA, Irwin MR, Olmstead R, Greendale G. Yoga for persistent fatigue in breast cancer survivors: a randomized controlled trial. Cancer. 2012 Aug 1;118(15):3766-75. doi: 10.1002/cncr.26702. Epub 2011 Dec 16. PMID 22180393
- [Background] Cramer H, Lauche R, Klose P, Lange S, Langhorst J, Dobos GJ. Yoga for improving health-related quality of life, mental health and cancer-related symptoms in women diagnosed with breast cancer. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD010802. doi: 10.1002/14651858.CD010802.pub2. PMID 28045199
- [Background] Stone PC, Minton O. Cancer-related fatigue. Eur J Cancer. 2008 May;44(8):1097-104. doi: 10.1016/j.ejca.2008.02.037. Epub 2008 Apr 1. PMID 18381237
- [Background] Johnson JA, Garland SN, Carlson LE, Savard J, Simpson JSA, Ancoli-Israel S, Campbell TS. Bright light therapy improves cancer-related fatigue in cancer survivors: a randomized controlled trial. J Cancer Surviv. 2018 Apr;12(2):206-215. doi: 10.1007/s11764-017-0659-3. Epub 2017 Nov 10. PMID 29127575
- [Background] Zhang Y, Lin L, Li H, Hu Y, Tian L. Effects of acupuncture on cancer-related fatigue: a meta-analysis. Support Care Cancer. 2018 Feb;26(2):415-425. doi: 10.1007/s00520-017-3955-6. Epub 2017 Nov 11. PMID 29128952
- [Background] Kampshoff CS, van Dongen JM, van Mechelen W, Schep G, Vreugdenhil A, Twisk JWR, Bosmans JE, Brug J, Chinapaw MJM, Buffart LM. Long-term effectiveness and cost-effectiveness of high versus low-to-moderate intensity resistance and endurance exercise interventions among cancer survivors. J Cancer Surviv. 2018 Jun;12(3):417-429. doi: 10.1007/s11764-018-0681-0. Epub 2018 Mar 1. PMID 29497963
- [Background] Group BRAH: The Behavioral Health Crisis: A Road Map for Academic Health Center Leadership in Healing Our Nation, in http://whsc.emory.edu/blueridge/publications/archive/Blue%20Ridge%202019-2020-FINAL.pdf (ed): Accessed Oct 2020, 2019
- [Background] Hernandez-Reif M, Field T, Ironson G, Beutler J, Vera Y, Hurley J, Fletcher MA, Schanberg S, Kuhn C, Fraser M. Natural killer cells and lymphocytes increase in women with breast cancer following massage therapy. Int J Neurosci. 2005 Apr;115(4):495-510. doi: 10.1080/00207450590523080. PMID 15809216
- [Background] Hernandez-Reif M, Ironson G, Field T, Hurley J, Katz G, Diego M, Weiss S, Fletcher MA, Schanberg S, Kuhn C, Burman I. Breast cancer patients have improved immune and neuroendocrine functions following massage therapy. J Psychosom Res. 2004 Jul;57(1):45-52. doi: 10.1016/S0022-3999(03)00500-2. PMID 15256294
- [Background] Jane SW, Wilkie DJ, Gallucci BB, Beaton RD. Systematic review of massage intervention for adult patients with cancer: a methodological perspective. Cancer Nurs. 2008 Nov-Dec;31(6):E24-35. doi: 10.1097/01.NCC.0000339242.51291.85. PMID 18987505
- [Background] Krohn M, Listing M, Tjahjono G, Reisshauer A, Peters E, Klapp BF, Rauchfuss M. Depression, mood, stress, and Th1/Th2 immune balance in primary breast cancer patients undergoing classical massage therapy. Support Care Cancer. 2011 Sep;19(9):1303-11. doi: 10.1007/s00520-010-0946-2. Epub 2010 Jul 20. PMID 20644965
- [Background] Kutner JS, Smith MC, Corbin L, Hemphill L, Benton K, Mellis BK, Beaty B, Felton S, Yamashita TE, Bryant LL, Fairclough DL. Massage therapy versus simple touch to improve pain and mood in patients with advanced cancer: a randomized trial. Ann Intern Med. 2008 Sep 16;149(6):369-79. doi: 10.7326/0003-4819-149-6-200809160-00003. PMID 18794556
- [Background] Listing M, Krohn M, Liezmann C, Kim I, Reisshauer A, Peters E, Klapp BF, Rauchfuss M. The efficacy of classical massage on stress perception and cortisol following primary treatment of breast cancer. Arch Womens Ment Health. 2010 Apr;13(2):165-73. doi: 10.1007/s00737-009-0143-9. Epub 2010 Feb 19. PMID 20169378
- [Background] Wilkinson S, Barnes K, Storey L. Massage for symptom relief in patients with cancer: systematic review. J Adv Nurs. 2008 Sep;63(5):430-9. doi: 10.1111/j.1365-2648.2008.04712.x. PMID 18727744
- [Background] Qin S, Xiao Y, Chi Z, Zhu D, Cheng P, Yu T, Li H, Jiao L. Effectiveness and safety of massage in the treatment of anxiety and depression in patients with cancer: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Sep 25;99(39):e22262. doi: 10.1097/MD.0000000000022262. PMID 32991424
- [Background] Fink J, Burns J, Perez Moreno AC, Kram JJF, Armstrong M, Chopp S, Maul SJ, Conway N. A Quality Brief of an Oncological Multisite Massage and Acupuncture Therapy Program to Improve Cancer-Related Outcomes. J Altern Complement Med. 2020 Sep;26(9):820-824. doi: 10.1089/acm.2019.0371. PMID 32924553
- [Background] Greenlee H, DuPont-Reyes MJ, Balneaves LG, Carlson LE, Cohen MR, Deng G, Johnson JA, Mumber M, Seely D, Zick SM, Boyce LM, Tripathy D. Clinical practice guidelines on the evidence-based use of integrative therapies during and after breast cancer treatment. CA Cancer J Clin. 2017 May 6;67(3):194-232. doi: 10.3322/caac.21397. Epub 2017 Apr 24. PMID 28436999
- [Background] Listing M, Reisshauer A, Krohn M, Voigt B, Tjahono G, Becker J, Klapp BF, Rauchfuss M. Massage therapy reduces physical discomfort and improves mood disturbances in women with breast cancer. Psychooncology. 2009 Dec;18(12):1290-9. doi: 10.1002/pon.1508. PMID 19189275
- [Background] Billhult A, Lindholm C, Gunnarsson R, Stener-Victorin E. The effect of massage on immune function and stress in women with breast cancer--a randomized controlled trial. Auton Neurosci. 2009 Oct 5;150(1-2):111-5. doi: 10.1016/j.autneu.2009.03.010. Epub 2009 Apr 18. PMID 19376750
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Diaz-Rodriguez L, Cuesta-Vargas AI, Fernandez-Delas-Penas C, Arroyo-Morales M. Attitudes towards massage modify effects of manual therapy in breast cancer survivors: a randomised clinical trial with crossover design. Eur J Cancer Care (Engl). 2012 Mar;21(2):233-41. doi: 10.1111/j.1365-2354.2011.01306.x. Epub 2011 Nov 8. PMID 22060159
- [Background] Mustian KM, Roscoe JA, Palesh OG, Sprod LK, Heckler CE, Peppone LJ, Usuki KY, Ling MN, Brasacchio RA, Morrow GR. Polarity Therapy for cancer-related fatigue in patients with breast cancer receiving radiation therapy: a randomized controlled pilot study. Integr Cancer Ther. 2011 Mar;10(1):27-37. doi: 10.1177/1534735410397044. Epub 2011 Mar 7. PMID 21382958
- [Background] Pan YQ, Yang KH, Wang YL, Zhang LP, Liang HQ. Massage interventions and treatment-related side effects of breast cancer: a systematic review and meta-analysis. Int J Clin Oncol. 2014 Oct;19(5):829-41. doi: 10.1007/s10147-013-0635-5. Epub 2013 Nov 26. PMID 24275985
- [Background] Kinkead B, Schettler PJ, Larson ER, Carroll D, Sharenko M, Nettles J, Edwards SA, Miller AH, Torres MA, Dunlop BW, Rakofsky JJ, Rapaport MH. Massage therapy decreases cancer-related fatigue: Results from a randomized early phase trial. Cancer. 2018 Feb 1;124(3):546-554. doi: 10.1002/cncr.31064. Epub 2017 Oct 17. PMID 29044466
- [Background] Ironson G, Field T, Scafidi F, Hashimoto M, Kumar M, Kumar A, Price A, Goncalves A, Burman I, Tetenman C, Patarca R, Fletcher MA. Massage therapy is associated with enhancement of the immune system's cytotoxic capacity. Int J Neurosci. 1996 Feb;84(1-4):205-17. doi: 10.3109/00207459608987266. PMID 8707483
- [Background] Diego MA, Field T, Hernandez-Reif M, Shaw K, Friedman L, Ironson G. HIV adolescents show improved immune function following massage therapy. Int J Neurosci. 2001 Jan;106(1-2):35-45. doi: 10.3109/00207450109149736. PMID 11264907
- [Background] Shor-Posner G, Miguez MJ, Hernandez-Reif M, Perez-Then E, Fletcher M. Massage treatment in HIV-1 infected Dominican children: a preliminary report on the efficacy of massage therapy to preserve the immune system in children without antiretroviral medication. J Altern Complement Med. 2004 Dec;10(6):1093-5. doi: 10.1089/acm.2004.10.1093. PMID 15674006
- [Background] Rapaport MH, Schettler P, Breese C. A preliminary study of the effects of a single session of Swedish massage on hypothalamic-pituitary-adrenal and immune function in normal individuals. J Altern Complement Med. 2010 Oct;16(10):1079-88. doi: 10.1089/acm.2009.0634. PMID 20809811
- [Background] Rapaport MH, Schettler P, Bresee C. A preliminary study of the effects of repeated massage on hypothalamic-pituitary-adrenal and immune function in healthy individuals: a study of mechanisms of action and dosage. J Altern Complement Med. 2012 Aug;18(8):789-97. doi: 10.1089/acm.2011.0071. Epub 2012 Jul 9. PMID 22775448
- [Background] Donoyama N, Ohkoshi N. Effects of traditional Japanese massage therapy on gene expression: preliminary study. J Altern Complement Med. 2011 Jun;17(6):553-5. doi: 10.1089/acm.2010.0209. Epub 2011 May 19. PMID 21595543
- [Background] Loft P, Petrie KJ, Booth RJ, Thomas MG, Robinson E, Vedhara K. Effects of massage on antibody responses after hepatitis B vaccination. Psychosom Med. 2012 Nov-Dec;74(9):982-7. doi: 10.1097/PSY.0b013e31826fb7d2. Epub 2012 Oct 15. PMID 23071344
- [Background] Best TM, Gharaibeh B, Huard J. Stem cells, angiogenesis and muscle healing: a potential role in massage therapies? Br J Sports Med. 2013 Jun;47(9):556-60. doi: 10.1136/bjsports-2012-091685. Epub 2012 Nov 29. PMID 23197410
- [Background] Kalauokalani D, Cherkin DC, Sherman KJ, Koepsell TD, Deyo RA. Lessons from a trial of acupuncture and massage for low back pain: patient expectations and treatment effects. Spine (Phila Pa 1976). 2001 Jul 1;26(13):1418-24. doi: 10.1097/00007632-200107010-00005. PMID 11458142
- [Background] Licciardone JC, Russo DP. Blinding protocols, treatment credibility, and expectancy: methodologic issues in clinical trials of osteopathic manipulative treatment. J Am Osteopath Assoc. 2006 Aug;106(8):457-63. PMID 16943515
- [Background] Myers SS, Phillips RS, Davis RB, Cherkin DC, Legedza A, Kaptchuk TJ, Hrbek A, Buring JE, Post D, Connelly MT, Eisenberg DM. Patient expectations as predictors of outcome in patients with acute low back pain. J Gen Intern Med. 2008 Feb;23(2):148-53. doi: 10.1007/s11606-007-0460-5. Epub 2007 Dec 8. PMID 18066631
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009